CLINICAL TRIAL: NCT03333642
Title: Ileal Interposition With Sleeve Gastrectomy for Type 2 Diabetes Mellitus Treatment
Brief Title: Surgery Treatment of Type 2 Diabetes Mellitus Patients With Grade 1 Obesity and Overweight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Federal de Bonsucesso (Other)
Responsible Party: Principal Investigator, Leonardo Rocha Ferraz, Surgeon MD, Hospital Federal de Bonsucesso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67955917.2.0000.5253
Record Dates: First submitted 2017-10-23; First posted 2017-11-07 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus; Obesity; Overweight
Keywords: diabetes; metabolic surgery; ileal interposition
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duodenal Ileal interposition (Experimental): Duodenal Ileal Interposition with Sleeve Gastrectomy.
  Interventions: Procedure: Duodenal Ileal Interposition with Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Duodenal Ileal Interposition with Sleeve Gastrectomy — Laparoscopic or open Duodenal Ileal Interposition with Sleeve Gastrectomy

SUMMARY:
This study evaluate the Duodenal Ileal Interposition with Sleeve Gastrectomy for Type 2 Diabetes Mellitus in grade 1 obesity and overweight patients.

DETAILED DESCRIPTION:
A clinical trial, 1-arm treatment (Duodenal Ileal Interposition with Sleeve Gastrectomy for Type 2 Diabetes Mellitus), including 50 research subjects with type 2 diabetes mellitus and obesity class I or overweight. The main objective is to analyse the effect on glycemic control after 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of type 2 diabetes mellitus;
* Patients of both sexes treated with oral antidiabetic agents and / or insulins,
* Stable antidiabetic medication in the last 8 weeks prior to selection, if the therapy includes insulin, the mean daily dose should not have been changed by more than 10% in the last 8 weeks;
* HbA1c> 7.0%;
* Age> 20 years and <65 years;
* Body mass index (BMI) of 25 to 35 kg / m²;
* Agree to sign the consent form;

Exclusion Criteria:

* Diabetes mellitus type 1 (anti-glutamic acid decarboxylase(GAD) positive) or anti-GAD negative body with low β-cell function (peptide C after stimulation <0.5 ng / ml);
* Recent vascular event (myocardial infarction, coronary angioplasty or encephalic vascular accident in the last 6 months);
* Malignant neoplasm;
* Portal hypertension;
* Difficulty to cooperate with segment;
* Low ability to understand surgery;
* Unrealistic expectations of results;
* Cognitive deficit;
* Current pregnancy;
* Moderate or severe mood disorder; severe anxiety; eating disorders (based on Substance-Related Disorders DSM-V criteria);
* Chemical dependence or alcoholism (based on Substance-Related Disorders DSM-V criteria).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Remission of type 2 Diabetes at 24 months | 2 years
  Number of patients with glycated hemoglobin (HbA1c) of 6.0% or less, without use of diabetes medications

SECONDARY OUTCOMES:
Control of type 2 diabetes | 2 years
  Number of patients with glycated hemoglobin (HbA1c) < 6.5%, but still in use of oral anti diabetic drugs and/or insulin

OTHER OUTCOMES:
Quality of life assessment | Before and 1, 3, 6, 12, 18 and 24 months after surgery
  Application of World Health Organization's Quality of Life questionnaire (WHOQOL-BREF)
Measurement of surgical adverse events | 2 years
  Use of Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo R Ferraz, MD, Principal Investigator — Hospital Federal de Bonsucesso
Locations (1):
- Hospital Federal de Bonsucesso, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided